CLINICAL TRIAL: NCT05142150
Title: Palliation in Gynae-oncology: Patients Expectations and Assessment of Care
Brief Title: Palliation in Gynae-oncology: Patients Expectations and Assessment of Care (PEACE)
Acronym: PEACE
Status: Recruiting | Type: Observational
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: Australia New Zealand Gynaecological Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: GCIG SB-001/NSGO-CTU-PEACE
Record Dates: First submitted 2021-10-08; First posted 2021-12-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Gynaecological Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — Hematology/ biochemistry: haemoglobin, white blood cell ( WBC) Count, neutrophils, platelets, albumin, C-Reactive protein (CRP), lactate dehydrogenase (LDH), alkaline phosphatase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patient satisfaction with end of life care. Questionnaire to be completed at baseline and every 8 week.
  Interventions: Other: Questionaire
- Carer: Carer satisfaction with care leading up to the time of death and the quality of the patient's death. Questionnaire to be completed at baseline and every 8 weeks,and 5-7 weeks after patient deceased.
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — Patient questionaires collecting data on quality of life, illness management, communication and decision making. Patient report data of end of life care ( i.e administration of chemotherapy, surgical interventions, palliative care involvement, hospital admissions) through as self reported diary.
  Carer for patients questionnaires their satisfaction with care. 5-7 weeks after patient deceased carer completes bereavement questionnaire and quality of death and dying.

SUMMARY:
The overall aim is to assess the feasibility and acceptability of collecting data on the patients and carers perception of care as well as to prospectively monitor end of life care.

DETAILED DESCRIPTION:
Prospective observational cohort study.

Little is known about end of life care (EOL) in patients with ovarian or other gynaecological cancers. Patients typically have a high symptom burden and following several prior lines of therapy or the development of platinum resistant disease response rates to further active treatment are limited. Eliciting patients' values and preferences for end-of-life care and shared decision-making are central elements of patient-centered EOL care. The aim of this study is to assess the feasibility of collecting data on patient satisfaction towards end of life. Preliminary data on patient and carer satisfaction with care, the importance of aspects of care, as well as end of life treatment will also be collected. The study will also assess the carer satisfaction with care during bereavement and with the patient's dying experience.

The study will recruit beyond the targeted number of 73 patients number if the study is progressing favourably. Ideally, each patient will nominate a carer to also complete questionnaires and the carer will be able to assist in completing the diary, although this is not mandatory.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion only if all of the following criteria are fulfilled:

1. Patients with any advanced gynecological malignancy and a life expectancy of approximately 4 months as estimated by their treating physician*. Potential patient groups include, but are not limited to, those with platinum-resistant/refractory recurrent epithelial ovarian cancer (PRR-EOC), metastatic/recurrent cervical or endometrial cancer progressing after platinum-based chemotherapy; high grade/undifferentiated metastatic uterine sarcoma progressing after first-line chemotherapy etc.
2. Patients may be on active cancer treatment, about to commence active cancer treatment or under observation/palliative care.
3. Age ≥ 18 years
4. Able (both physically and cognitively) to complete patient-reported outcome measures independently in languages that are available in this study (i.e. without assistance from hospital translator).

Exclusion Criteria:

A patient will not be eligible for inclusion if any of the following criteria are fulfilled:

1. Unable to be comply with the protocol.
2. A medical or psychological condition that limits the patient´s capacity to give informed consent, such as cognitive impairment, delirium, psychosis etc.
3. Participation in another clinical trial.

A patient will be asked to appoint a carer.

Inclusion criteria carer:

1. Age ≥ 18 years
2. A relative or close friend who is actively supporting the patient in her illness
3. Able (both physically and cognitively) to complete questionnaires independently in languages that are available in this study (i.e. without assistance from hospital translator).

Exclusion criteria carer

A carer will not be eligible for inclusion if any of the following criteria are fulfilled:

1. Unable to be comply with the protocol
2. A medical or psychological condition that limits the carer´s capacity to give informed consent, such as cognitive impairment, delirium, psychosis etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in end of life with advanced gynaecological malignancies and their carers.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who complete scheduled assessments with Canadian Health Care Evaluation Project (CANHELP) instrument, CANHELP Lite Individualised version | Within 42 days before their death
  To study the feasibility of collecting data on patient satisfaction with care. In all CANHELP Lite versions response options for each item range from 1'not at all satisfied' to 5 'completely satisfied'. All versions have an overall satisfaction with care score, as well as scores on each of the individual domains. All scores are re-scaled to range between 0 (worst possible value) to 100 (best possible value).

SECONDARY OUTCOMES:
Number of carers who complete scheduled assessments with Canadian Health Care Evaluation Project (CANHELP) Lite Individualized Caregiver | Within 42 days before patient's death
  To study the feasibility of collecting data on carer satisfaction with care. In all CANHELP Lite versions response options for each item range from 1'not at all satisfied' to 5 'completely satisfied'. All versions have an overall satisfaction with care score, as well as scores on each of the individual domains. All scores are re-scaled to range between 0 (worst possible value) to 100 (best possible value).
Number of carers who complete scheduled assessments with Canadian Health Care Evaluation Project (CANHELP) Lite bereavement and Quality of Death and Dying (QODD) questionnaire | Within 42 days of death up to 5-7 weeks after patient deceased.
  To study the feasibility of collecting data on carer satisfaction with care leading up to the time of death and the quality of the patient´s death. CANHELP response options range from 1'not at all satisfied' to 5 'completely satisfied', with an overall satisfaction with care score and scores on each individual domains. All scores are re-scaled to range 0 (worst possible value) to 100 (best possible value). The QODD questionnaire has 24 items that assess aspects of dying and death. The QODD questionnaire contains 14 additional items that assess cargiver's demographic characteristics and relation to the deceased. Response options for each item are rated on a scale from 0 (terrible) to 10 (almost perfect). The items provide a single score, derived as a mean of the item values, transformed to a 0 to 100 scale.
Number of patients who received chemotherapy and other interventions as well as palliative care | Within 42 days before their death
  To study use of chemotherapy, surgical interventions as well as palliative care involvement
Patient satisfaction with care | Baseline up to 5-7 weeks after patient deceased
  Patient satisfaction will be assessed with CANHELP Lite Individualized. In all CANHELP Lite versions response options for each item range from 1'not at all satisfied' to 5 'completely satisfied' . A 'not applicable/not discussed' response option for items that patients/cares felt was not relevant to their situation. All versions have an overall satisfaction with care score, as well as scores on each of the individual domains. All scores are re-scaled to range between 0 (worst possible value) to 100 (best possible value). The questionnaires will be administered and scored in accordance with the user manual.
Carers satisfaction with care | Baseline up to 5-7 weeks after patient deceased
  Satisfaction will be assessed with CANHELP Lite bereavement and quality of death and dying (QODD) questionnaire.
  The QODD questionnaire has 24 items that assess various aspects of dying and death including whether the patient's symptoms were adequately controlled, whether dignity was maintained, time spent with loved ones in days leading up to death and whether the patient's wishes were adhered to. The QODD questionnaire also contains 14 additional items that assess the cargiver's demographic characteristics and relation to the deceased. The response options for each item are rated on a scale from 0 (terrible) to 10 (almost perfect). The items provide a single score, derived as a mean of the item values, transformed to a 0 to 100 scale.
The importance of aspects of care for patients | Baseline up to 5-7 weeks after patient deceased
  Importance of aspects of care will be assessed through CANHELP Lite.
The importance of aspects of care for carers | Baseline up to 5-7 weeks after patient deceased
  Importance of aspects of care assessed through CANHELP Lite.

CONTACTS AND LOCATIONS:
Locations (1):
- The Norwegian Radium Hospital, Oslo, Norway